CLINICAL TRIAL: NCT04407572
Title: Zinc Vitamin D and b12 Levels in the Covid-19 Positive Pregnant Women
Brief Title: Evaluation of the Relationship Between Zinc Vitamin D and b12 Levels in the Covid-19 Positive Pregnant Women
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Ayşegül Bestel (Unknown); İbrahim Polat (Unknown); Merve Aldıkaçtıoğlu Talmaç (Unknown)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: zinc-dvit-covid19
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: COVID; Zinc Deficiency; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum zinc, vitamin d vitamin b12 levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Serum zinc, vitamin d vitamin b12 levels . — Serum zinc, vitamin d vitamin b12 levels of 45 patients will be measured and evaluated together with the information of the patients.

SUMMARY:
Zinc d vitamin and b12 serum levels in covid-19 positive pregnants will be compared in terms of patients' responses to computed tomography and treatment.

DETAILED DESCRIPTION:
Serum zinc, vitamin d vitamin b12 levels of 45 patients will be measured and evaluated together with the information of the patients.

ELIGIBILITY:
Inclusion Criteria:

* covid-19 positive pregnant women
* under 18 or more than 45 years old

Exclusion Criteria:

* vitamin D , Vitamin B12 or Zinc supplement use
* Multivitamine use
* have taken vitamin supplements in the past 3 months
* use of medicines for vitamin deficiency
* having metabolic disease covid-19 negative pregnant women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women between 18-45 years old with positive covid-19 pcr test results
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Serum zinc, vitamin d vitamin b12 deficiency levels | 2 months
  Serum zinc, vitamin d vitamin b12 levels of 45 patients will be measured and evaluated together with the information of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes